CLINICAL TRIAL: NCT01065857
Title: Phase III, Multicenter, Randomized, Assessor-blind Study to Evaluate the Safety and Efficacy of CitraFleet (Sodium Picosulphate) as an Evacuating Treatment Prior to Colonoscopy.
Brief Title: Safety and Efficacy Study of CitraFleet (Sodium Picosulphate) as an Evacuating Treatment Prior to Colonoscopy.
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Laboratorios Casen-Fleet S.L.U. (Industry)
Collaborators: Trial Form Support S.L. (Other); Apices Soluciones S.L. (Industry)
Responsible Party: Ángel Navarro Lima, M.D. / European Medical Affairs Director, Laboratorios Casen-Fleet S.L.U.
Allocation: Randomized | Model: Parallel | Masking: Single
Other Study IDs: CF-PICOS2006
Record Dates: First submitted 2010-02-08; First posted 2010-02-09 (Estimated); Last update posted 2011-04-15 (Estimated); Status verified 2011-04

CONDITIONS: Subjects Undergoing a Complete Exploratory Diagnostic Colonoscopy for the First Time.
Keywords: Colonoscopy, Preparation, Evacuating, Bowel Cleansing.
MeSH Terms: interventions — picosulfate sodium; Polyethylene Glycols; Sodium Bicarbonate

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- Citrafleet (Experimental): The day prior to the colonoscopy in two dose times, first at 15:00h and second at 20:00h.
  Interventions: Drug: Sodium picosulphate, light magnesium oxide and anhydride citric acid.
- Klean Prep (Active Comparator): The day prior to the colonoscopy from 16:00h to 20:00h.
  Interventions: Drug: Polyethylene glycol, KCl, NaCl, sodium sulphate anhydrous and sodium bicarbonate.
- Citrafleet Exploratory (Experimental): The day of the colonoscopy in two dose times, first at 06:00h and second at 09:00h.
  Interventions: Drug: Sodium picosulphate, light magnesium oxide and anhydride citric acid.

INTERVENTIONS:
Drug: Sodium picosulphate, light magnesium oxide and anhydride citric acid. — 2 Single-dose sachets containing sodium picosulphate (0.01g/sachet), light magnesium oxide (3.50g/sachet) and anhydrous citric acid (10.97g/sachet).
  Other Names: Citrafleet
  Arms: Citrafleet; Citrafleet Exploratory
Drug: Polyethylene glycol, KCl, NaCl, sodium sulphate anhydrous and sodium bicarbonate. — 4 sachets containing Polyethylene glycol 3350 (59 gr), KCl (0.7425 gr), NaCl (1.465 gr), sodium sulphate anhydrous (5.685 gr), sodium bicarbonate (1.685 gr).
  Other Names: KleanPrep PEG 4l
  Arms: Klean Prep

SUMMARY:
The purpose of this study is to determine any significant differences in the efficacy and acceptability between CitraFleet and Klean Prep® (polyethylene glycol) for the preparation of gastrointestinal subjects undergoing a colon examination.

DETAILED DESCRIPTION:
The composite principal objective of the current study will therefore be, to determine any significant differences in the joint variable of efficacy and acceptability between CitraFleet and Klean Prep® (polyethylene glycol) for the preparation of subjects undergoing a colon examination.

The evaluation will be carried out by two blinded assessors, independent of the investigator who performed the procedure (endoscopist investigator). It will be assessed from images of different sections of the colon: cecum, ascending, transverse, descending and rectum and subsequent confirmation by Principal Investigator if an agreement has been reached between the two blinded assessors or whether it is necessary to reach consensus.

The evaluation of the subject's acceptability will be assessed using a 5 point scale which assesses the difficulty of taking the product, the degree of discomfort caused by it, and the taste of the drug.

The secondary objective is to evaluate the safety of CitraFleet.

In addition a second exploratory arm of CitraFleet was included in this study (CitraFleet Exploratory arm). The study is not powered to make formal statistical comparisons for this arm. Exploratory assessment of this arm against the main CitraFleet regimen and Klean-Prep will be made in order to run future trials design with this schedule.

ELIGIBILITY:
Inclusion Criteria:

* Subjects who are between 18 and 80 years of age.
* Subjects undergoing complete colonoscopy and therefore require prior preparation with either Klean Prep® or CitraFleet.
* Subjects capable of maintaining appropriate oral hydration during the intestinal preparation process.
* Subjects that have provided written informed consent.
* Subjects in whom the use of any of the study drugs (KleanPrep®,CitraFleet) is not contraindicated.
* Subjects who can communicate with the study personnel and comply with study requirements.
* Subjects undergoing a complete exploratory diagnostic colonoscopy for the first time.

Exclusion Criteria:

* Severe renal insufficiency.
* Ascites.
* Congestive heart failure.
* Gastrointestinal obstruction, gastric retention, intestinal perforation and/or ileus.
* Megacolon and/or toxic colitis.
* Nausea and/or vomiting and/or abdominal pain.
* Severe dehydration.
* Hypermagnesemia.
* Rhabdomyolysis.
* Pregnant women.
* Subjects who have participated in a clinical trial in the previous 30 days.
* Abdominal surgery for any acute process (for example acute appendicitis).
* Active inflammatory intestinal disease.
* Known allergy to any of the active ingredients or excipients of the study drugs.
* Subjects not providing written informed consent.
* Subjects not complying with all of the inclusion criteria.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 547 (Estimated)
Dates: Start 2010-01; Primary Completion 2010-06 (Actual); Study Completion 2011-02 (Actual)

PRIMARY OUTCOMES:
Percentage of subjects that achieve 'excellent' or 'good' cleansing in the Fleet® Grading Scale for Bowel Cleansing. | 24 hours
Percentage of subjects who find the agent easy to take or tolerable using a 5 point scale which assesses, the difficulty of taking the product, the degree of discomfort caused by it, and the taste of the drug, recorded in the subject questionnaire | 24 hours

SECONDARY OUTCOMES:
Frequency of adverse reactions. | 24 hours

CONTACTS AND LOCATIONS:
Overall Officials: Miguel A. Muñoz-Navas, M.D., Principal Investigator — Clínica Universitaria de Navarra
Locations (15):
- Spain (15):
  - H. Universitari Vall´d Hebron, Barcelona, Barcelona
  - H. Clínic, Barcelona, Barcelona
  - H. General Universitario Reina Sofía, Córdoba, Córdoba
  - H. Universitario Virgen de las Nieves, Granada, Granada
  - H. General Universitario Gregorio Marañón, Madrid, Madrid
  - H. Universitario Puerta de Hierro, Madrid, Madrid
  - H. Infanta Elena, Valdemoro, Madrid
  - H. Universitario Virgen de la Arrixaca, Murcia, Murcia
  - H. Regional Universitario Carlos Haya, Málaga, Málaga
  - Clínica Universitaria de Navarra, Pamplona, Navarre
  - H. Universitario Central de Asturias, Oviedo, Oviedo
  - H. Virgen Macarena, Seville, Sevilla
  - H. Universitario de Canarias, San Cristóbal de La Laguna, Tenerife
  - H. Universitario La Fé, Valencia, Valencia
  - H. Basurto, Bilbao, Vizcaya